CLINICAL TRIAL: NCT01829217
Title: A Phase II Trial of Sunitinib in Never-smokers With Lung Adenocarcinoma: Identification of Oncogenic Alterations Underlying Sunitinib Sensitivity
Brief Title: Sunitinib in Never-Smokers With Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Geoffrey Oxnard, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-086
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): 42 day cycle, taken orally every day for the first 28 days followed by 14 days off
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied. It also means that the FDA has not yet approved sunitinib for your type of cancer.

Sunitinib has been approved by the FDA for treatment of gastrointestinal stromal tumors, advanced renal cell carcinoma and advanced pancreatic neuroendocrine tumors. While most chemotherapies work by interfering with cancer cell replication, sunitinib works by blocking certain protein signals within the cell. Because sunitinib works differently from standard intravenous chemotherapies, we call it a "targeted therapy." This drug has also been used in other research studies and information from those other research studies suggests that this agent may help to slow the growth of some NSCLC tumors.

In this research study, we are looking to see if sunitinib may stop certain NSCLC tumors from growing. The study focuses on a type of NSCLC, adenocarcinoma, which has previously been found to be more sensitive to other kinds of oral targeted therapies. This study will focus specifically on (1) adenocarcinoma tumors that do not carry a mutation in a known cancer gene (EGFR, KRAS, or ALK) and occur in patients that never smoked (less than 100 cigarettes in their lifetime) or (2) adenocarcinoma tumors that have a mutation in the RET gene.

DETAILED DESCRIPTION:
Primary Objectives

- To evaluate the objective response rate (ORR) to sunitinib in never-smokers with lung cancers that are wild-type for EGFR, KRAS, and ALK in a single-arm phase II trial

Secondary Objectives

* To identify oncogenic alterations underlying sensitivity to sunitinib through performing nextgeneration sequencing (NGS) of lung cancers treated with sunitinib
* To explore the activity of sunitinib in lung cancers known to harbor a RET rearrangements and other genomic alterations in targets of sunitinib (e.g. cKIT, PDGFRa, PDGFRb).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced (stage IV or recurrent) non-small cell lung cancer
* Adenocarcinoma histology of any variant, including adenosquamous histology
* Wild-type for mutations in EGFR, KRAS and ALK
* Must have < 100 cigarettes smoked lifetime OR known to harbor a RET rearrangement OR another potentially targetable genomic alteration as defined per protocol
* Disease must be measureable per RECIST 1.1
* At least one prior systemic therapy (adjuvant or palliative)
* 18 years or older
* Life expectancy of greater than 4 weeks
* Adequate ECOG performance status 0 or 1
* Adequate organ function as defined in the protocol
* Adequate tumor tissue for the correlative analyses on study, or must undergo a biopsy to obtain adequate tissue

Exclusion Criteria:

* Pregnant or breastfeeding
* Chemotherapy within 4 weeks of entering study, or lack of recover from adverse events to grade 1 or less due to systemic agents administered more than 4 weeks earlier
* Radiation therapy within 2 weeks prior to entering study
* Major surgery within 4 weeks prior to entering the study
* Receiving any other investigational agents
* Known untreated, symptomatic or progressive brain metastases; presence of carcinomatous meningitis; history of intracranial hemorrhage or brain metastases requiring chronic steroids
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib
* Use of certain inhibitors and inducers of CYP3A4
* Grade 3 or 4 hemoptysis or hemorrhage within 4 weeks prior to study entry
* History of significant bleeding disorder unrelated to cancer
* Poorly controlled hypertension
* Severe cardiovascular disease
* Prolongation of corrected QT interval
* History of a different malignancy except: cervical cancer in situ, basal or squamous cell carcinoma of the skin, low risk centralized prostate cancer
* HIV positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Oxnard, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Cooper AJ, Kobayashi Y, Kim D, Clifford SE, Kravets S, Dahlberg SE, Chambers ES, Li J, Rangachari D, Nguyen T, Costa DB, Rabin MS, Wagle N, Sholl LM, Janne PA, Oxnard GR. Identification of a RAS-activating TMEM87A-RASGRF1 Fusion in an Exceptional Responder to Sunitinib with Non-Small Cell Lung Cancer. Clin Cancer Res. 2020 Aug 1;26(15):4072-4079. doi: 10.1158/1078-0432.CCR-20-0397. Epub 2020 Apr 20. PMID 32312893
- [Derived] Wu H, Shih JY, Yang JC. Rapid Response to Sunitinib in a Patient with Lung Adenocarcinoma Harboring KIF5B-RET Fusion Gene. J Thorac Oncol. 2015 Sep;10(9):e95-e96. doi: 10.1097/JTO.0000000000000611. No abstract available. PMID 26291023

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: 42 day cycle, taken orally every day for the first 28 days followed by 14 days off
  Sunitinib
Period: Overall Study
Arm/Group | Sunitinib
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 67 [53 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of patients with evidence of complete or partial response per RECIST1.1 criteria.
Time Frame: ORR was assessed at 6 weeks post-registration and every 6 weeks until date of documented disease progression or death, up to January 23, 2017 (approximately 44 months).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 13
percentage of participants | 7.69 [0.22 to 36.05]

ADVERSE EVENTS:
Time Frame: Adverse events should be reported from start of study intervention through 30 days after the last dose of study treatment. AEs were assessed through January 23, 2017, approximately 44 months.
Description: Because this drug is commercially available, only grade 3 adverse events are reported here.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 7/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=13)
Anemia (Blood and lymphatic system disorders) | 2 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 (4)
Palpitations (Cardiac disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (3)
Eye pain (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 5 (10)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (11)
Nausea (Gastrointestinal disorders) | 6 (9)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (7)
Edema limbs (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Fatigue (General disorders) | 9 (20)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (3)
Mucosal infection (Infections and infestations) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 3 (8)
Weight loss (Investigations) | 2 (4)
White blood cell decreased (Investigations) | 5 (11)
Anorexia (Metabolism and nutrition disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (8)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (5)

LIMITATIONS AND CAVEATS:
This study was closed to accrual due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT01829217/Prot_SAP_000.pdf